CLINICAL TRIAL: NCT04726046
Title: Prospective Randomized Control Study of Clinical Effectiveness of Prophylactic Antibiotics Therapy in Laparoscopic Cholecystectomy on Infection Rate
Brief Title: Effectiveness of Prophylactic Antibiotics Therapy in Laparoscopic Cholecystectomy on Infection Rate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ChonbukNUH
Record Dates: First submitted 2017-09-18; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2017-09

CONDITIONS: Cholecystitis
Keywords: GB stone
MeSH Terms: conditions — Cholecystitis | interventions — Cefotetan

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic treatment group (Experimental): They were Antibiotic treatment group (AG, cefotetan 1g, 1 dose/prophylactic) before surgery.
  Interventions: Drug: Cefotetan
- Non-antibiotic treatment group (No Intervention): They were Non-antibiotics treatment such as cefotetan 1g before surgery.

INTERVENTIONS:
Drug: Cefotetan — Cefotetan (as Disodium) 1 GM Injection before surgery
  Other Names: antibiotics group
  Arms: Antibiotic treatment group

SUMMARY:
529 patients performed elective LCC at Chonbuk National University Hospital between April 2014 and August 2015. Total 509 patients were enrolled by inclusion criteria.

They were randomized studied by comparing with antibiotic group (n=249, AG, cefotetan 1g, 1 dose/prophylactic) and non-antibiotic group (n=260, NAG) by table of random numbers. The clinical variables were pre and post-operatively blood tests enclude WBC, ESR, CRP, body temperatures, symptoms and imaging of chest x-ray to evaluate the infections.

DETAILED DESCRIPTION:
529 patients performed elective LCC at Chonbuk National University Hospital between April 2014 and August 2015. Total 509 patients were enrolled by inclusion criteria. They were randomized studied by comparing with antibiotic group (n=249, AG, cefotetan 1g, 1 dose/prophylactic) and non-antibiotic group (n=260, NAG) by table of random numbers. The clinical variables were pre and post-operatively blood tests enclude WBC, ESR, CRP, body temperatures, symptoms and imaging of chest x-ray to evaluate the infections.

ELIGIBILITY:
Inclusion Criteria:

patients who have diagnosed -cholecystitis with / without GB stone, GB polyp

Exclusion Criteria:

1. Suspected cholangitis and GB cancer
2. CBD stone history
3. Preoperative administration of antibiotics within 7days.
4. Suspected pregnancy
5. Open conversion.
6. Patients refuse this study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
surgical complication | 30days
  surgical site infection

CONTACTS AND LOCATIONS:
Overall Officials: Jae Do Yang, Study Director — Chonkbuk national university

IPD SHARING:
Plan to Share IPD: No